CLINICAL TRIAL: NCT03820154
Title: A Bridging Study Investigating the Diagnostic Equivalence of the SPT Tape in Comparison With the Conventional SPT Using ALK SoluprickR Allergen Extracts in Patients With Inhalation Allergy
Brief Title: Diagnostic Equivalence of the Skin Prick Test Tape vs. Conventional Skin PrickTest
Acronym: SPTTapeD1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Prof. Dr. Claus Bachert BVBA (Individual)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CBauchert
Record Dates: First submitted 2018-09-23; First posted 2019-01-29 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Allergic Rhinitis; Allergic Asthma; Allergic Conjunctivitis; Food Allergy
MeSH Terms: conditions — Rhinitis, Allergic; Conjunctivitis, Allergic; Food Hypersensitivity | interventions — Patch Tests

STUDY DESIGN:
Intervention Model Description: Comparison of conventional Skin Prick Test vs. Tape SPT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Skin Prick Test TAPE (Active Comparator): The Skin Prick Test Tape is an innovative sterile "all-in" drug carrying 8 allergens and 2 control solutions including prick needles in one Tape for easy use and standardization. Single use. Reading of wheal reactions after 15 minutes, facilitated by stripes with the allergen names.
  Interventions: Diagnostic Test: Skin Prick Test TAPE
- Skin Prick Test (Active Comparator): The conventional SPT is the world-wide standard in allergy Type 1 diagnosis for inhalant and food allergens. Drops of allergens are applied to the forearm and, with the help of a lancet, brought into the skin. Reading of wheal reactions after 15 minutes.
  Interventions: Diagnostic Test: Skin Prick Test

INTERVENTIONS:
Diagnostic Test: Skin Prick Test — Skin Prick Testing with inhalant allergens
  Arms: Skin Prick Test
Diagnostic Test: Skin Prick Test TAPE — Skin Prick Testing with a Tape, integrating the allergens and needles
  Arms: Skin Prick Test TAPE

SUMMARY:
Testing of a new ready-to-use Tape in comparison to the currently used skin prick test for the diagnosis of allergies. Assessment of clinical equivalence of the SPT Tape for representative common inhalant allergens to conventional SPT in terms of wheal reaction positivity and overall safety. Tests are performed in patients who have a medical history of relevant allergic rhinitis to any of the tested allergens.

DETAILED DESCRIPTION:
An open-label, single site bridging study. Subjects with a history of in-halation allergies will be tested in parallel with the SPT Tape and with the conventional SPT procedure using one forearm each.

In each patient, a panel of 8 allergens with the SPT Tape and with the conventional SPT is applied on the two forearms one time only.

The following Soluprick® allergens and control solutions will be evaluated:

Positive control, negative control, Phleum pratense, birch, Dermatophagoides pteronyssinus, D. farinae, dog dander, cat dander, mugwort, Alternaria sp. The allergens used for the SPT and the SPT Tape are identical Soluprick allergen solutions; allergens will be applied in the same location and order on both arms.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be included only, if

  1. they were informed about the nature, meaning, and scope of the study, and if they provided written consent to their participation
  2. they are at least 18 years of age,
  3. they have a history of allergic rhinitis due to grass and/or birch pollen, house dust mites, mugwort, cat and/or dog dander, and/or Alternaria since 2 years or more

Exclusion Criteria:

* Subjects may not be included, if

  1. they are impaired in understanding nature, meaning, and the scope of the study, or are incapable of giving written informed consent,
  2. they suffer from diseases, show other conditions, or take medications, which might impact the skin tests or might contradict the correct conduct and evaluation of the study. In particular this includes the following:

     1. acute allergy,
     2. history of systemic reactions or hypersensitivity to allergens, abuse of drugs or alcohol
     3. severe diseases,
     4. impaired reactivity of the skin (e.g. hyperkeratosis, ichthyosis, urticaria factitia) and acute chronic eczema in the skin test areas, skin infections,
     5. pregnancy or nursing,
     6. treatment with β-blockers,
     7. treatment with antihistamines or systemic glucocorticoids during the last 4 weeks, with astemizol during the last 12 weeks,
     8. treatment with tricyclic antidepressants benzodiazepines, and neuroleptic drugs which may have histamine-antagonistic effects during the last 2 weeks,
     9. participation in any other medication study at the study time

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2019-03-31 (Estimated); Study Completion 2019-07-30 (Estimated)

PRIMARY OUTCOMES:
Wheal diameters | 15 min
  Maximal wheal diameter in millimeter

SECONDARY OUTCOMES:
Visual Analogue Scale on Comfort | 30 min
  Visual Analogue Scale from 0-10 cm from "not at all unpleasant" to "very unpleasant"
Patient' s preference | 30 min
  Patients are asked to select the test they would prefer

CONTACTS AND LOCATIONS:
Overall Officials: Martin Wagenmann, MD, Principal Investigator — University pf Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: No